CLINICAL TRIAL: NCT04606901
Title: Comparison of Time to Full Recovery From Muscle Paralysis (TOF>0.9) and Extubation Using Sugammadex Versus Neostigmine/Glycopyrrolate in Patients With Pulmonary Disease in the Outpatient Bronchoscopy Suite
Brief Title: Comparison of Time to Extubation Using Sugammadex or Neostigmine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 26881
Record Dates: First submitted 2020-10-13; First posted 2020-10-28 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Neuromuscular Blockade; Chronic Obstructive Pulmonary Disease
Keywords: Nondepolarizing neuromuscular blockade; sugammadex; bronchoscopy; outpatient; lung disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Neostigmine; Glycopyrrolate; Sugammadex

STUDY DESIGN:
Intervention Model Description: Study groups will be treated equally except for delivery of the neuromuscular blockade reversal medication
Who Masked: Participant, Investigator
Masking Description: Medications will be provided by Merck, Sharp & Dohme Corp and will be delivered to the inpatient pharmacy in such a way as to blind the pharmacist. Patients will also not know which medication they are receiving
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex (Active Comparator): Patients in this arm of the study will receive Sugammadex as the drug used to reverse neuromuscular blockade.
  Interventions: Drug: sugammadex
- Neostigmine/Glycopyrrolate (Active Comparator): Patients in this arm of the study will receive Neostigmine/Glycopyrrolate as the drugs used to reverse neuromuscular blockade
  Interventions: Drug: neostigmine/glycopyrrolate

INTERVENTIONS:
Drug: neostigmine/glycopyrrolate — neuromuscular blockade reversal agents
  Other Names: prostigmin/robinul
  Arms: Neostigmine/Glycopyrrolate
Drug: sugammadex — neuromuscular blockade reversal agent
  Other Names: Bridion
  Arms: Sugammadex

SUMMARY:
A prospective blinded randomized clinical trial to compare time to extubation using Sugammadex versus Neostigmine/glycopyrrolate as reversal agents after use of neuromuscular blockade agents in an outpatient bronchoscopy suite.

DETAILED DESCRIPTION:
This research study will have the design of a blinded randomized clinical trial. The pharmacist will be blinded to the study medication given. The anesthesia provider cannot be blinded because he/she will need to determine the proper dose and timing of the neuromuscular blocker reversal medication (the study medications) given at the end of the procedure. The study will recruit 80 patients coming to Temple University Hospital for an outpatient bronchoscopy biopsy procedure that requires general anesthesia with neuromuscular blockade. Rocuronium will be the neuromuscular blockade medication given in this study. Inclusion criteria for these patients will include those age >18 who have a diagnosis of chronic obstructive pulmonary disease (COPD) and/or idiopathic lung disease (ILD) and who require medical treatment for the same; these patients will have American society of anesthesiology physical status (ASA PS) 3-4 based on their pulmonary disease alone.The patients will then be randomly assigned to one of two study arms (40 per arm). Patients in one arm of the study will receive Sugammadex and patients in the other arm will receive neostigmine/glycopyrrolate for reversal of neuromuscular blockade. Due to the nature of bronchoscopy for biopsy, the depth of anesthesia at the end of the case will be difficult to predict; the length of the cases may vary some (although most will be approximately one hour), and patients' metabolism of neuromuscular blocking agents is very much dependent on their personal medication regimens and liver function. Each patient's depth of neuromuscular blockade will be followed using the TwitchView monitor, a commercially available, an electromyography (EMG) based monitor. The TwitchView measures muscle response to delivered electrical stimuli (2Hz) which are sent in sets of 4X0.5 seconds apart (most commonly). The muscles controlled by the ulnar nerve will be followed during this study. Return of muscle strength after reversal agents are given is considered complete when the ratio of the strength of the response to the fourth electrical stimulus to the first stimulus is 0.9. Multiple time points will be recorded, including train of four measurement (TOF) every 5 minutes during the procedure, time and TOF at the end of the procedure, time of reversal medication dosing, time of TOF>0.9 and time of extubation. Reversal medication will be given as soon as each patient's procedure is complete and the patient meets appropriate criteria for reversal for each respective medication. Comparison of the data from the two arms of the study will then be made.

ELIGIBILITY:
Inclusion Criteria:

1. has diagnosis of COPD or ILD
2. ASA 3 or 4
3. procedure requires general anesthesia in the outpatient bronchoscopy suite
4. glomerular filtration rate > 30 ml/min

Exclusion Criteria:

1. pregnant women
2. prisoners
3. those unable to consent for themselves
4. procedures not requiring general anesthesia
5. ASA 1 or 2

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Hauck, DO PhD, Principal Investigator — Lewis Katz School of Medicine at Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Only deidentified data from the study will be made available to other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Started | 28 | 30
Completed | 28 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (8.7) | 65.0 (8.8) | 65.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 18 | 23 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 11 | 7 | 18
  White | 15 | 19 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Minutes to Return of Baseline Muscle Tone
Description: number of minutes from reversal dose to Train of Four (TOF) >0.9 indicating full reversal of neuromuscular blockade agent
Time Frame: 1-20 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 28 | 30
minutes | 3.9 (2.0) | 12.9 (9.8)

2. Secondary Outcome: Number of Minutes to Extubation
Description: number of minutes from Train of Four (TOF) >0.9 to extubation of the patient
Time Frame: 1-30 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 28 | 30
minutes | 11.9 (8.3) | 17.7 (10.5)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected over the entire period of the study. 2 years and 3 months.
Description: The clinicaltrials.gov definition for Adverse Events or Serious Adverse Events was followed for this study. The definition can be found below:
  Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT04606901/Prot_SAP_001.pdf